CLINICAL TRIAL: NCT03391752
Title: More-2-Eat Phase 2: Spread/Scaling up Improved Nutrition Care to Detect and Treat Hospital Malnutrition.
Brief Title: More-2-Eat Phase 2: Scaling and Spread of the Integrated Nutrition Pathway for Acute Care
Status: Completed | Type: Observational
Sponsor: University of Waterloo (Other)
Collaborators: Canadian Malnutrition Task Force (Other); Canadian Frailty Network (Other)
Responsible Party: Principal Investigator, Heather Keller, Schlegel-University of Waterloo Research Chair, Nutrition & Aging, University of Waterloo
Other Study IDs: KT2017-01
Record Dates: First submitted 2018-01-01; First posted 2018-01-05 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Malnutrition
Keywords: malnutrition, screening, assessment, treatment
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Royal Alexandria: Administrative records
  Interventions: Combination Product: Integrated Nutrition Pathway for Acute Care
- Pasqua Regional hospital: Administrative records
  Interventions: Combination Product: Integrated Nutrition Pathway for Acute Care
- Concordia Hospital: Administrative records
  Interventions: Combination Product: Integrated Nutrition Pathway for Acute Care
- Niagara General Hospital: Administrative records
  Interventions: Combination Product: Integrated Nutrition Pathway for Acute Care
- Hospital 6: Administrative Records
  Interventions: Combination Product: Integrated Nutrition Pathway for Acute Care
- Hospital 7: Administrative Records
  Interventions: Combination Product: Integrated Nutrition Pathway for Acute Care
- Hospital 8: Administrative Records
  Interventions: Combination Product: Integrated Nutrition Pathway for Acute Care
- Hospital 9: Administrative Records
  Interventions: Combination Product: Integrated Nutrition Pathway for Acute Care
- Hospital 10: Administrative records
  Interventions: Combination Product: Integrated Nutrition Pathway for Acute Care

INTERVENTIONS:
Combination Product: Integrated Nutrition Pathway for Acute Care — algorithm to guide care processes with respect to nutrition e.g. screening on admission, diagnosis with subjective global assessment, early treatment with medication pass of oral nutritional supplement

SUMMARY:
More-2-Eat Phase 2 provides the opportunity to extend the implementation of the Integrated Nutrition Pathway to a total of 10 hospitals and more than 20 medical/surgical units. Building on the success of More-2-Eat Phase 1, key components of this implementation study will be a registry for self-managed data entry and reports and a community of practice to support implementation of nutrition screening at admission to hospital, subjective global assessment to diagnose and triage patients to care pathways and medication pass of a small amount of nutrient dense oral nutritional supplement. Success with implementation and impact on key patient outcomes will be determined.

DETAILED DESCRIPTION:
Malnutrition in hospital patients is a growing problem, with 20-45% of patients already malnourished at admission. As 70% of malnourished patients are also frail, early detection and treatment of malnutrition is one way to improve the outcomes of frail older adults. To improve the detection and treatment of these conditions, the PI developed the Integrated Nutrition Pathway for Acute Care (INPAC) that guides hospital staff on when to conduct key nutrition care activities to improve outcomes (e.g. screening at admission).

In More-2-Eat (April 2015-March 2017), 5 Canadian hospital units in 4 provinces received funding to implement INPAC. Each hospital, with support from a research team had 1 year to implement INPAC. All 5 hospitals were successful in improving detection and treatment of malnutrition, and started to screen for frailty. Clinical care was transformed in the study units; for example all sites progressed from low baseline or no screening at admission to a rate of 75%. Findings also demonstrate improvement in clinical outcomes such as a shorter length of stay. An online INPAC Implementation Toolkit was developed to promote mobilization of this knowledge. What is not known is whether or not the results can be replicated under normal circumstances (i.e., no external funding for implementation at a hospital site).

To sustain and expand on this success, a Phase 2 knowledge translation project is proposed that will involve the five original Phase 1 sites and five further hospitals as Phase 2 sites. The goal of the second phase is to see if Phase 1 sites can spread success to other units within their hospitals and if Phase 2 sites can achieve similar results across a broader group of patients.

The end product will be a sustainable model including a community of practice supported by our partner the Canadian Malnutrition Task Force, and a self-serve registry that allows sites to collect and report data to change their practice. Investigators will also confirm capacity of INPAC activities to improve clinical outcomes across diverse settings. This knowledge translation and implementation study will demonstrate the potential to transform clinical nutrition care, benefiting all pre-frail and frail older adults.

ELIGIBILITY:
Inclusion Criteria:

* Patient on the study unit

Exclusion Criteria:

* patients not on the study unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients admitted to study units in one of the 10 hospitals included will be subject to the improved nutrition care processes; those that are malnourished will be offered a variety of treatments including medication pass
Sampling Method: Non-Probability Sample
Enrollment: 5158 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
success with implementation | 19 months
  rates of screening, diagnosis and treatment with medication pass per month of the study

SECONDARY OUTCOMES:
Adverse events while in hospital (fall, new infection etc.) | 19 months
Length of stay | 19 months
  Average length of stay for patients admitted to the study unit; monthly average
Readmission rate | 19 months
  number of patients per month discharged and readmitted to the hospital within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Heather Keller, PhD, Principal Investigator — University of Waterloo
Locations (9):
- Canada (9):
  - Royal Alexander Hospital, Edmonton, Alberta
  - Brandon Regional Health Centre, Brandon, Manitoba
  - Concordia Hospital, Winnipeg, Manitoba
  - Victoria General Hospital, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Lennox Addington County General Hospital, Napanee, Ontario
  - Niagara Health Systems, Niagara Falls, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Pasqua Hospital, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
UWSpace at the University of Waterloo
Supporting Information: Analytic Code
Time Frame: 2020

REFERENCES:
- [Derived] Laur C, Bell J, Valaitis R, Ray S, Keller H. The role of trained champions in sustaining and spreading nutrition care improvements in hospital: qualitative interviews following an implementation study. BMJ Nutr Prev Health. 2021 Sep 28;4(2):435-446. doi: 10.1136/bmjnph-2021-000281. eCollection 2021. PMID 35028514